CLINICAL TRIAL: NCT07122128
Title: Saliva as Early Detection Tool for Oral Cancer
Brief Title: EVALUATION OF SALIVA AS LIQUID BIOPSY FOR EARLY DETECTION OF ORAL CANCER IN PATIENTS WITH ORAL-SUBMUCOUS FIBROSIS (OSMF)
Acronym: Sal
Status: Recruiting | Type: Observational
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Sindh Higher Education Commission (Unknown)
Responsible Party: Principal Investigator, Prof. Binafsha Manzoor Syed, Professor, Liaquat University of Medical & Health Sciences
Other Study IDs: SalivaP01; Sal001 (Other: Liaquat University of Medical and Health Sciences)
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: The Study Focuses on the Saliva as Potential Source of Early Detection of Oral Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal healthy volunteers: oral examination will be done, those without any oral infection, oral submucous fibrosis or cancer will be included in health volunteer group
  Interventions: Diagnostic Test: saliva a a diagnostic tool for early detection of oral cancer
- oral submucous fibrosis: Patients with oral submucous fibrosis both with and without limited mouth opening
  Interventions: Diagnostic Test: saliva a a diagnostic tool for early detection of oral cancer
- oral cancer patients: patients with biopsy proven oral cancer
  Interventions: Diagnostic Test: saliva a a diagnostic tool for early detection of oral cancer

INTERVENTIONS:
Diagnostic Test: saliva a a diagnostic tool for early detection of oral cancer — Three groups will be compared on the basis of cytology, genes and biochemical analysis

SUMMARY:
Oral cancer is the top cancer in Pakistan, accounting for 27%, and it has a high mortality rate due to late-stage diagnosis. It primarily affects the lips, tongue, cheeks, and floor of the mouth. Major risk factor for oral cancer development is pan supari chhaliya chewing.

Patients often develop a pre-malignant condition, oral submucous fibrosis, resulting in limited mouth opening. Thus, patients are diagnosed at an advanced level and poor survival. Therefore, saliva appears a potential mode of evaluation for early detection. This project aims to evaluate salivary cells, genes and biochemistry of the saliva among health volunteers and compare it with that of the patients with oral submucous fibrosis and oral cancer.

DETAILED DESCRIPTION:
The project aims to evaluate salivary cytology, genes and biochemistry of the healthy normal population and compare it with that of the oral submucous fibrosis and oral cancer. For salivary experiments 3 cc of fresh saliva will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* patients with oral submucous fibrosis
* patients with biopsy proven oral cancer

Exclusion Criteria:

* patients with oral infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The three groups will be recruited: healthy volunteers with unremarkable oral examination, patients with oral submucous fibrosis regardless of mouth opening and biopsy proven oral cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
salivary cytology | 1 year
  A method will be developed for evaluation of detection of oral cancer
evaluation of telomere length of salivary cells | 1 year
  Telomere length will be evaluation in the saliva of three groups
evaluation of biochemicals of saliva | 1 year
  saliva of three groups will be compared on the basis of salivary enzymes

OTHER OUTCOMES:
A scoring system will be developed for the screening of patients at risk of oral submucous fibrosis | 2 years
  A scoring system will be developed including cytology, genetic and biochemistry and algorithm will be designed for accurate assessment of the oral cancer

CONTACTS AND LOCATIONS:
Overall Officials: Binafsha Manzoor Prof. Syed, PhD, Principal Investigator — Liaquat University of Medical and Health Sciences
Locations (1):
- Medical Research Center, Jāmshoro, Sinch, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD includes: Group, age, gender, smoking status, oral hygiene status, saliva collection date, salivary cytology parameters, telomere length, p53 status